CLINICAL TRIAL: NCT00933907
Title: Study Title: Study for Dermatological Evaluation of Topic Compatibility Primary and Accumulated Dermical Irritability and Dermical Sensitivity for the Product Dermacyd PH_DESILSTY_FR (Lactic Acid) .
Brief Title: Dermacyd PH_DESILSTY_FR (Lactic Acid) - Compatibility - Stay on Frutal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACAC_L_04807
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Hygiene

ARMS (1):
- Dermacyd PH_DESILSTY_FR (Lactic Acid) (Experimental): Dermacyd PH_DESILSTY_FR (Lactic Acid) sample will be applied like a curative. Physiologic solution and mineral oil will be also used as a control sample.
  Interventions: Drug: LACTIC ACID(ND)

INTERVENTIONS:
Drug: LACTIC ACID(ND) — Treatment duration: 6 weeks

SUMMARY:
Primary Objective:

To demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd PHDESILSTYFR.

ELIGIBILITY:
Inclusion criteria:

* Phototype Skin I,II, III e IV Integral skin test in the region
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion;

Exclusion criteria:

* Lactation or gestation
* Use of Antiinflammatory 30 days and/or immunossupression drugs for until 3 months before volunteers selection
* Disease which can cause immunosuppresion, such as diabetes, HIV
* Personnel history of atopy
* History of sensitivity or irritation for topic products
* Cutaneous active disease (local and/or general) which can modify the study results
* Use of new drugs and/or cosmetics during the study
* Cutaneous reactive
* Previous participation in studies using the same product in test
* Volunteer which has immunodeficiency congenital or acquired
* Relevant history or confirmation of alcohol or other drugs abuse
* Intolerance detected or suspected for some component of the sample tested
* Medecin or sponsor employees or their close family.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the absence of primary and accumulated dermical irritability and dermical sensitivity by using International Contact Dermatitis Research Group (ICDRG) scale. | From the treatment start to the end of the study( treatment period 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil